CLINICAL TRIAL: NCT07360678
Title: Comparing the Garmin Venu 3 for Non-Invasive Vital Sign Monitoring to a Hospital-Grade Monitor
Acronym: GARMIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, David Ruttens, Prof. Dr., Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Z-2025082; CIV-25-07-053536 (Other: EUDAMED)
Record Dates: First submitted 2025-09-22; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Validation of Vital Signs Measured by a Consumer-grade Smartwatch
Keywords: Vital signs; Garmin; Accuracy; Heart rate; Respiratory rate; Peripheral Oxygen Saturation (SpO2)

STUDY DESIGN:
Intervention Model Description: Each participant will be continuously monitored for a minimum of one full night and up to a maximum of 24 hours using both a hospital-grade monitor (Philips IntelliVue X2) and a Garmin Venu 3 smartwatch. Recruitment will take place within the pneumology ward. Upon completion of the monitoring period, participants will be asked to complete the Smartwatch Rating Scale (SRS) questionnaire to assess their experience with the smartwatch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients admitted to the pulmonology ward (Experimental): Patients admitted to the pulmonology ward of Ziekenhuis Oost-Limburg, Genk, Belgium.
  Interventions: Device: Garmin Venu 3 + Philips Intellivue X2; Other: Smartwatch rating scale questionnaire

INTERVENTIONS:
Device: Garmin Venu 3 + Philips Intellivue X2 — Each participant will be continuously monitored for a minimum of one full night and up to a maximum of 24 hours using both a hospital-grade monitor (Philips IntelliVue X2) and a Garmin Venu 3 smartwatch.
Other: Smartwatch rating scale questionnaire — Upon completion of the monitoring period, participants will be asked to complete the Smartwatch Rating Scale (SRS) questionnaire

SUMMARY:
This clinical trial evaluates the accuracy of the Garmin Venu 3 smartwatch in measuring vital signs (heart rate, respiratory rate, SpO₂) compared to the clinically validated Philips IntelliVue X2. The study aims to determine whether the consumer-grade smartwatch can provide reliable data for remote patient monitoring, early hospital discharge, and chronic disease management, offering a more accessible and affordable alternative to MDR-certified devices.

DETAILED DESCRIPTION:
Wearable technology has rapidly evolved from fitness tracking tools to potential clinical-grade devices capable of non-invasive monitoring of vital signs. Among these, smartwatches equipped with optical sensors and accelerometers now offer continuous measurements of parameters such as heart rate, respiratory rate, and blood oxygen saturation (SpO2). The Garmin Venu 3 represents a new generation of commercially available smartwatches that provide vital sign monitoring outside of controlled medical environments.

Despite their growing popularity and technological advancements, the clinical validity of smartwatches remains unknown. Applying for medical device regulation (MDR) certification is a long and expensive process, something not all companies can or want to invest in. Besides, the devices that are MDR certified are often very expensive, something not possible to use in an average patient population without extensive funding. For the use of (non-MDR certified) smartwatches into clinical workflows or remote patient monitoring systems, these devices must demonstrate accuracy and reliability comparable to gold-standard hospital-grade monitors.

The Philips IntelliVue X2 is a widely used and clinically validated multi-parameter patient monitoring system employed in acute care setting. It provides high-fidelity, real-time monitoring of vital signs and serves as an appropriate benchmark for evaluating the performance of customer-grade devices.

Comparing measurements obtained with the Garmin Venu 3 against the IntelliVue X2 is essential to determine whether the smartwatch can serve as a reliable tool for continuous vital sign tracking in real-world clinical scenarios. This is particularly relevant for use cases such as early hospital discharge, remote patient monitoring and chronic disease management where accessibility, affordability, convenience and user compliance are critical.

This clinical trial seeks to assess the agreement and accuracy of the Garmin Venu 3 in measuring key physiological parameters such as heart rate, respiratory rate, and SpO2 compared to the Philips Intellivue X2 in a diverse patient population. Demonstrating clinical equivalence or acceptable accuracy margins would support the potential use of the Garmin Venu 3 in remote or supplemental monitoring roles within modern (hybrid) healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent
* Adults older than 18 years of age
* Speak and understand the Dutch language
* Hospitalized for at least another 24 hours

Exclusion Criteria:

* Life expectancy is less than 30 days
* Patient is isolated due to infection control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean absolute difference between the Garmin Venu 3 and a hospital-grade monitor in measuring heart rate up to 24 hours. | From enrollment to the end of treatment at 24 hours
  For heart rate, the mean absolute difference will be calulated between the measurements performed with the Garmin Venu 3 and the measurements performed with the Philips Intellivue X2
Mean absolute difference between the Garmin Venu 3 and a hospital-grade monitor in measuring respiratory rate up to 24 hours. | From enrollment to the end of treatment at 24 hours
  For respiratory rate, the mean absolute difference will be calculated between the measurements performed with the Garmin Venu 3 and the measurements performed with the Philips IntelliVue X2
Mean absolute difference between the Garmin Venu 3 and a hospital-grade monitor in measuring peripheral oxygen saturation up to 24 hours. | From enrollment to the end of treatment at 24 hours
  For peripheral oxygen satuation (SpO2), the mean absolute difference will be calculated between the measurements performed with the Garmin Venu 3 and the measurements performed with the Philips IntelliVue X2.

SECONDARY OUTCOMES:
User experience of the Garmin Venu 3 as measured by the Smartwatch Rating Scale | From enrollment to the end of treatment at 24 hours
  User experience of the Garmin Venu 3 as measured by the Smartwatch Rating Scale
Number of artefacts during measurements performed when the participant is awake vs measurements performed when the participant is asleep (expressed in % measurements) | From enrollment to the end of treatment at 24 hours
  Measurements reported as a '0' due to the inability of the device to perform a correct measurement will be labeled as false.
Time to detection of a sudden drop in SpO2 or clinical deterioration measured by the Garmin Venu 3 vs a hospital-grade monitor | From enrollment to the end of treatment at 24 hours
  In the event of patient deterioration, changes may be reflected in SpO2 levels. This endpoint will evaluate the time taken by the Garmin Venu 3 compared to a hospital-grade monitor to detect such changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Raw data regarding the vital parameter measurements with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code